CLINICAL TRIAL: NCT04030299
Title: Longitudinal Outcomes of Over-the-Counter Hearing Aids
Brief Title: Longitudinal Outcomes of Hearing Aids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yu-Hsiang Wu (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, Yu-Hsiang Wu, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 201905847; R01DC015997-01A1 (NIH)
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Presbycusis
Keywords: Presbycusis; Hearing aid
MeSH Terms: conditions — Presbycusis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- OTC Group (Experimental): In this group, the over-the-counter fitting will be used to provide hearing aids.
  Interventions: Device: Over-the-counter fitting

INTERVENTIONS:
Device: Over-the-counter fitting — In this group, pre-configured hearing aids, which simulate over-the-counter hearing aids, will be provided to subjects. Subjects will take the full initiative and responsibility for learning and using hearing aids.

SUMMARY:
Age-related hearing loss is a substantial national problem due to its high prevalence and significant psychosocial consequences. Although hearing aids (HAs) are the primary intervention for the management of age-related hearing loss, only 15-30% of those who could benefit from HAs actually seek them out. HA adoption rates are even worse for people with lower income and for racial and ethnic minorities. One of the most commonly reported reasons for people not seeking HA intervention is the high cost of HAs and the associated audiological fitting services. Because HAs fitted using the audiologist-based service-delivery model are unaffordable, more and more Americans (1.5 million in 2010) purchase amplification devices via over-the-counter (OTC) service-delivery models to compensate for their impaired hearing.

Although OTC amplification devices are gaining popularity and are regarded as an important option for promoting accessible and affordable hearing healthcare, it is unclear if they are viable solutions for age-related hearing loss as OTC models exclude professional services. Further, although there is some evidence supporting the effectiveness of OTC HAs, all previous studies measured short-term outcomes (e.g., 6 weeks). It is unknown what the long-term outcomes of OTC HAs would look like. The outcomes could improve across time because users may eventually figure out how to use HAs. On the other hand, the outcomes of OTC HAs could become poorer across time because, unlike traditional HA fitting, users do not have professionals to support them. Therefore, the overall goal of this project is to examine the longitudinal changes in OTC HA outcomes over 3 months.

DETAILED DESCRIPTION:
Although hearing aids (HAs) are the first treatment of choice for age-related hearing loss, only 15-30% of those older Americans who could benefit, actually seek HAs out and use them. HA adoption rates are even lower for people with lower income and for racial and ethnic minorities. Although the answer to why so few older adults seek or use amplification is multidimensional, one common thread is that many people believe that HAs fitted using the audiologist-based model cost too much. Therefore, it is not surprising that there has been increased advocacy for a variety of over-the-counter (OTC) service-delivery models, which have increasingly been identified as important options for managing mild-to-moderate age-related hearing loss.

Is the amplification intervention delivered using the OTC model an appropriate solution for age-related hearing loss? Although there is some evidence supporting the effectiveness of OTC HAs, all previous studies measured short-term outcomes (e.g., 6 weeks). It is unknown what the long-term outcomes of OTC HAs would look like. The purpose of this project is to examine the longitudinal changes in OTC HA outcomes over 3 months. Older adults with age-related hearing loss will be recruited. Pre-configured hearing aids (that simulate OTC hearing aids) will be provided to subjects. Subjects will take the full initiative and responsibility for learning and using hearing aids. HA outcomes will be measured at 6-week and 12-week post intervention.

ELIGIBILITY:
Inclusion Criteria:

* adult-onset, bilateral, mild-to-moderately severe sensorineural hearing loss

Exclusion Criteria:

* Non-native speaker of English

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsiang Wu, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
The proposed research will include data from a total of 45 participants with hearing loss recruited State of Iowa and surrounding areas. The final dataset will include laboratory data (e.g., speech recognition score) and self-reported demographic and behavioral data (e.g., questionnaire). Contact the principle investigator for data access.
Time Frame: The date will be available starting 6 months after publication of the main findings of the trial.
Access Criteria: Even though the final dataset will be stripped of identifiers prior to release for sharing, there remains the possibility of deductive disclosure of subjects with the survey data being collected. Thus, we will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate technologies; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Background] Donahue A, Dubno JR, Beck L. Guest editorial: accessible and affordable hearing health care for adults with mild to moderate hearing loss. Ear Hear. 2010 Feb;31(1):2-6. doi: 10.1097/AUD.0b013e3181cbc783. No abstract available. PMID 20040828
- [Background] Lin FR, Thorpe R, Gordon-Salant S, Ferrucci L. Hearing loss prevalence and risk factors among older adults in the United States. J Gerontol A Biol Sci Med Sci. 2011 May;66(5):582-90. doi: 10.1093/gerona/glr002. Epub 2011 Feb 27. PMID 21357188
- [Background] Humes LE, Rogers SE, Quigley TM, Main AK, Kinney DL, Herring C. The Effects of Service-Delivery Model and Purchase Price on Hearing-Aid Outcomes in Older Adults: A Randomized Double-Blind Placebo-Controlled Clinical Trial. Am J Audiol. 2017 Mar 1;26(1):53-79. doi: 10.1044/2017_AJA-16-0111. PMID 28252160
- [Background] Brody L, Wu YH, Stangl E. A Comparison of Personal Sound Amplification Products and Hearing Aids in Ecologically Relevant Test Environments. Am J Audiol. 2018 Dec 6;27(4):581-593. doi: 10.1044/2018_AJA-18-0027. PMID 30458521
- [Background] Takahashi G, Martinez CD, Beamer S, Bridges J, Noffsinger D, Sugiura K, Bratt GW, Williams DW. Subjective measures of hearing aid benefit and satisfaction in the NIDCD/VA follow-up study. J Am Acad Audiol. 2007 Apr;18(4):323-49. doi: 10.3766/jaaa.18.4.6. PMID 17580727
- [Background] Gopinath B, Schneider J, Hartley D, Teber E, McMahon CM, Leeder SR, Mitchell P. Incidence and predictors of hearing aid use and ownership among older adults with hearing loss. Ann Epidemiol. 2011 Jul;21(7):497-506. doi: 10.1016/j.annepidem.2011.03.005. Epub 2011 Apr 21. PMID 21514179

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between September 2019 and September 2022. Participants were recruited from the an established participant registry and through mass emails to the University of Iowa community.
Period: Overall Study
Arm/Group | OTC Group
Started | 34
Completed | 24
Not Completed | 10
Not completed — Coronavirus disease 2019 (COVID-19) | 7
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | OTC Group
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.29 (7.68103)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Hearing Aid Benefit as Measured by the Glasgow Hearing Aid Benefit Profile (GHABP)
Description: The Glasgow Hearing Aid Benefit Profile (GHABP) is a questionnaire that measures hearing aid users' listening experience in four situations (TV listening, small conversation in quiet, conversation in noise, and group conversation). The score ranges from 0 (no benefit) to 5 (lots of benefit). The score at 1-week, 6-week and 12-week post intervention is the primary outcome.
Time Frame: 1-week, 6-week, and 12-week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OTC Group
Number analyzed (Participants) | 24
score on a scale
  1-week post-intervention | 3.68 (0.695)
  6-week post intervention | 3.55 (0.648)
  12-week post-intervention | 3.63 (0.715)

2. Secondary Outcome: Hearing Aid Performance/Benefit as Measured Using the Profile of Hearing Aid Performance (PHAP)
Description: The PHAP is a questionnaire designed to measures the performance of hearing aids in speech communication. The score ranges from 1 (good performance) to 99 (poor performance).
Time Frame: 1-week, 6-week, and 12-week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OTC Group
Number analyzed (Participants) | 24
score on a scale
  1-week post intervention | 30.5 (13.7)
  6-week post intervention | 30.4 (14.5)
  12-week post intervention | 29.5 (14.3)

3. Secondary Outcome: Hearing Handicap as Measured by Hearing Handicap Inventory for the Elderly (HHIE) or Hearing Handicap Inventory for Adults (HHIA)
Description: The HHIE and HHIA are questionnaires designed to measure subject's perceived hearing handicap. For subjects order and younger 65 years old, the HHIE and HHIA will be used, respectively. The score ranges from 0 (no handicap) to 100 (more handicap).
Time Frame: 1-week, 6-week, and 12-week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OTC Group
Number analyzed (Participants) | 22
score on a scale
  1-week post intervention | 20.2 (14.3)
  6-week post intervention | 13 (10.9)
  12-week post intervention | 17.7 (16.6)

4. Secondary Outcome: Hearing Aid Satisfaction as Measured by the Hearing Aid Satisfaction Survey (HASS)
Description: The HASS is a questionnaire developed to measures subject's perceived hearing aid satisfaction. The score ranges from 0 (low satisfaction) to 10 (high satisfaction).
Time Frame: 1-week, 6-week, and 12-week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OTC Group
Number analyzed (Participants) | 20
score on a scale
  1-week post intervention | 3.6 (0.66)
  6-week post intervention | 3.5 (0.63)
  12-week post intervention | 3.5 (0.73)

5. Secondary Outcome: Willingness-to-pay
Description: Willingness-to-pay (WTP) estimates the extent to which (in dollars) a subjects, at a maximum, is willing to pay out-of pocket for the amplification devices and the associated services used in the study..
Time Frame: 6-week and 12-week post intervention
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | OTC Group
Number analyzed (Participants) | 21
dollars
  6-week post intervention | 967.7 (1040)
  12-week post intervention | 1104.7 (1312)

6. Secondary Outcome: Quality of Life as Measured by the World Health Organization's Disability Assessment Schedule 2.0 (WHODAS 2.0)
Description: The WHODAS is a questionnaire designed to measure quality of life. The summary score ranges from 0 (No disability) to 100 (Full disability).
Time Frame: 1-week, 6-week, and 12-week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OTC Group
Number analyzed (Participants) | 24
score on a scale
  1-week post-intervention | 7.5 (7.1)
  6-week post-intervention | 6.7 (6.5)
  12-week post-intervention | 7.5 (7.0)

7. Secondary Outcome: Hearing Aid Satisfaction as Measured by the Satisfaction With Amplification in Daily Life (SADL)
Description: The SADL is a questionnaire designed to measures subject's perceived hearing aid satisfaction. The score ranges from 1 (low satisfaction) to 7 (high satisfaction).
Time Frame: 1-week, 6-week, and 12-week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OTC Group
Number analyzed (Participants) | 20
score on a scale
  1-week post intervention | 4.6 (1.3)
  6-week post intervention | 4.4 (1.2)
  12-week post intervention | 4.6 (1.4)

8. Secondary Outcome: Speech Recognition Performance as Measured by the Connected Speech Test (CST)
Description: The CST is a speech recognition test designed to simulate daily speech communication. The score ranges from 0 (understand no speech) to 100 (understand all speech).
Time Frame: 1-week, 6-week, and 12-week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OTC Group
Number analyzed (Participants) | 22
score on a scale
  1-week post intervention | 64.9 (27.8)
  6-week post intervention | 79.6 (13.5)
  12-week post intervention | 76.8 (17.1)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for each subject during their participation in the study, which averaged 12 weeks from the time the participants entered the study.
Arm/Group | OTC Group
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

LIMITATIONS AND CAVEATS:
Sample Size, ideal N would have been 34 but only 24 due to COVID-19. COVID-19 limited the acoustic environments subjects encountered. Homogeneity of sample in education level, socioeconomic status, and race.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT04030299/Prot_002.pdf
  • Informed Consent Form (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT04030299/ICF_000.pdf